CLINICAL TRIAL: NCT04208126
Title: Early Versus Late Initiation of ECMO Trial (ELIEO-Trial)
Brief Title: Early Versus Late Initiation of ECMO (Extracorporal Membrane Oxygenation) Trial (ELIEO-Trial)
Acronym: ELIEO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ELIEO
Record Dates: First submitted 2019-12-05; First posted 2019-12-23 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Acute Respiratory Distress Syndrome
Keywords: Acute Respiratory Distress Syndrome; Extracorporal membrane Oxygenation; Outcome; Ventilation Therapy; QOL
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Intervention Model Description: This trial is a prospective randomized multicenter trial that assigns patients to either a treatment for ARDS with an ECMO immediately after admission to the intensive care unit or conservative treatment.
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Early ECMO (Active Comparator): ECMO is placed immediately after admission to the intensive care unit
  Interventions: Device: ECMO
- Control (No Intervention): Conservative therapy unless failure of therapy.

INTERVENTIONS:
Device: ECMO — ECMO implantation immediately after ICU admission
  Arms: Early ECMO

SUMMARY:
This trial is a prospective randomized multicenter trial that assigns patients to either a treatment for Acute Respiratory Distress Syndrome (ARDS) with an Extracorporal Membrane Oxygenation (ECMO) immediately after admission to the intensive care unit or conservative treatment. The later can undergo ECMO following failure of conservative therapy as a rescue therapy. Patients will be included within 24 hours of the onset of symptoms of ARDS and will be randomized according to standard procedure. Follow-up will be performed until day 90 after study inclusion.

DETAILED DESCRIPTION:
Patients suffering acute ARDS defined according to the Berlin Definition starting from severe stage with acute onset and (i) ratio partial arterial pressure of oxygen fraction of inspired oxygen inspired oxygen fraction (PaO2/ FiO2) ≤ 200 (ii) Bilateral opacities consistent with pulmonary edema on frontal chest radiograph, and (iii) requirement for positive pressure ventilation via an endotracheal tube or non-invasive ventilation (iv) no clinical evidence of left atrial hypertension, or if measured, a Pulmonary Arterial Wedge Pressure (PAOP) less than or equal to 18 mm Hg (v) less than 96 hours from onset of ARDS (vi) less than 7 days from the initiation of mechanical ventilation will be treated by ECMO either within 24 hours to referral to an ARDS ECMO center or as rescue therapy after failure of conventional therapy.

Outcome measures have been chosen according to robustness and sensitivity to change. They are of high clinical impact and reflect the treatment effect desired by clinicians.

Primary efficacy endpoint: All cause mortality by 90-days.

Key secondary endpoints are:

2. 28 day all cause mortality 3. SOFA Organ Failure Scores at day at day 1-7, 14, 28 and 90 days 4. Duration of mechanical ventilation support 5. ICU length of stay

ELIGIBILITY:
Inclusion Criteria:

* ARDS as defined according to the Berlin Definition1
* The term "acute onset" is defined as follow: the duration of the hypoxemia criterion and the chest radiograph criterion must be ≤ 7 days at the time of randomization.
* Patients must be enrolled within 96 hours of onset of ARDS and no later than 7 days from the initiation of mechanical ventilation.

Exclusion Criteria:

* Age less than 18 years
* More than 7 days since initiation of mechanical ventilation
* more than 96 hours since meeting inclusion criteria
* patient, surrogate or physician not committed to full intensive care support
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 508 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2028-08 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
90 day all cause mortality | 90 days after study inclusion
  90 day all cause mortality

SECONDARY OUTCOMES:
Sepsis-related organ failure assessment score (SOFA) Organ Failure Scores | 1-14, 28 and 90 days after study inclusion
  SOFA Organ Failure Scores
Duration of mechanical ventilation | within 90 days after study inclusion
  Duration of mechanical ventilation
28 day all cause mortality | 28 days after study inclusion
  28 day all cause mortality
ICU length of stay | overall length of stay
  overall length of stay on ICU

CONTACTS AND LOCATIONS:
Overall Officials: Peter Rosenberger, Prof., Principal Investigator — University Hospital Tübingen
Locations (1):
- University hospital Tübingen, Tübingen, Germany